CLINICAL TRIAL: NCT07112820
Title: Contribution of Myocardial Perfusion Imaging in the Initial Assessment of Acute Coronary Syndromes Without ST Elevation for the Diagnosis of Myocardial Infarction or Differential Diagnoses
Acronym: APRICOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APRICOT
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Myocardial Infarction (MI)
Keywords: acute coronary syndrome without ST segment elevation; emergency cardiology
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: prospective single-centre cohort study for diagnostic purposes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: perfusion ultrasound — During the examination, the power of the probe will be increased in order to assess myocardial perfusion.
  The contrast agent bubbles are destroyed by applying a 'flash', i.e. a temporary increase in the power of the ultrasound beam. Systole after systole, on a recorded loop, the filling velocity of the myocardium, which depends on myocardial blood flow, is analysed. The assessment of perfusion is visual and qualitative.

SUMMARY:
Patients with myocardial infarction require invasive treatment involving coronary angiography to confirm the diagnosis and, in most cases, treatment by angioplasty/stenting. Trans-thoracic ultrasound is central to the initial management of patients admitted to hospital with acute coronary syndrome without ST segment elevation.

The aim of our study is therefore to compare perfusion ultrasound with coronary angiography and MRI in this population in order to determine whether the performance is satisfactory.

DETAILED DESCRIPTION:
Patients with myocardial infarction require invasive treatment via coronary angiography to confirm the diagnosis and, in most cases, treatment by angioplasty/stenting. In the case of acute coronary syndrome without ST segment elevation (NSTEMI), myocardial infarction is suspected but cannot be confirmed. The recommendations suggest that, in cases of low suspicion, a non-invasive ischaemia test should be performed, but in cases of high suspicion, coronary angiography should be performed immediately (1). In cases of NSTEMI, segmental kinetic abnormalities on echocardiography place the patient under high suspicion of infarction and justify coronary angiography without prior ischaemia testing. However, certain kinetic abnormalities may be related to causes other than infarction: stress cardiomyopathy (TakoTsubo), left bundle branch block, pacemaker stimulation, myocarditis, leading to unnecessary and potentially harmful invasive examinations. Transthoracic echocardiography (TTE) is central to the initial management of patients hospitalised for NSTEMI, both to confirm the diagnosis and to detect any immediate complications.The use of contrast agents during TEE is already recommended to improve the quality of the examination, as it increases the echogenicity of patients, and several studies have demonstrated its usefulness in analysing myocardial perfusion (2). The only contrast agent currently available in France is Sonovue® (Bracco Imaging). Microbubbles are lipid 'shells' containing a gas (sulphur), with a diameter similar to that of red blood cells (less than 7 μm). The behaviour of microbubbles in the circulation and capillaries can therefore be likened to that of red blood cells, which allows for better visualisation of all the structures through which blood flows (3). Its use is not contraindicated in the acute phase of a myocardial infarction and has few adverse effects (4).

Several studies have shown that the use of contrast agents during perfusion ultrasound can improve the diagnosis of ischaemic heart disease (5) and distinguish stress-induced heart disease (TakoTsubo) from myocardial infarction (6-8). No studies have looked at patients with kinetic disorders of other aetiologies (bundle branch block, pacemaker).

Furthermore, in certain patients presenting with actual myocardial infarction with segmental kinetic abnormalities but no significant coronary lesions on coronary angiography, myocardial MRI is of definite value in confirming or ruling out the diagnosis of healthy coronary artery infarction (1). However, the use of MRI in routine practice is severely limited by the lack of MRI facilities in many centres or by delays in obtaining results that are incompatible with the urgency of diagnosis.

Compared to computed tomography (CT) and MRI, the advantages of contrast-enhanced ultrasound are 1) the possibility of real-time imaging and 2) the absence of nephrotoxicity, risk of hyperthyroidism and radiation exposure. The aim of our study is therefore to compare perfusion ultrasound with coronary angiography and MRI in this population so that, if the results are satisfactory, certain invasive examinations currently considered essential can be avoided.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Hospitalised in cardiology as an emergency for acute coronary syndrome without ST segment elevation with indication for coronary angiography within 72 hours of admission
* Not yet undergone coronary angiography.
* Troponin >99th percentile, i.e. >27ng/l (troponin I, hypersensitive, Abbott)
* With de novo segmental kinetic disorder on TTE or ECG repolarisation disorder outside ST elevation
* Patient affiliated with a health insurance scheme
* French-speaking patient
* Patient who has given their free, informed and written consent

Exclusion Criteria:

Haemodynamically unstable patient: HR > 100 and/or systolic blood pressure < 90 mmHg and/or diastolic blood pressure < 60 mmHg and/or oxygen saturation < 92% in AA and/or clinical signs of hypoperfusion (mottling, cyanosis)

* Rhythmically unstable patient: sustained ventricular tachycardia, sudden death recovered.
* Patient with a known allergy to ultrasound contrast medium
* Patient with ST segment elevation.
* Patient with a contraindication to MRI.
* Patient with a caricatured picture of myocarditis (fever and/or significant biological inflammatory syndrome with CRP>50mg/l)
* Patients already included in a type 1 interventional research protocol (RIPH1)
* Patients under guardianship or curatorship
* Patients deprived of their liberty
* Patients under judicial protection
* Pregnant or breastfeeding patients (negative pregnancy test for women of childbearing age)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity (SE) and specificity (SP), positive predictive value (PPV) and negative predictive value (NPV) (diagnosis obtained by consensus of two cardiologists based on all blinded examinations of the ultrasound results). | inclusion visit
  Contrast-enhanced ultrasound (same measurements) according to recommendations, performed and interpreted by cardiologist 1, then reviewed and reinterpreted by the cardiologist.
  The reference diagnosis will be established by two cardiologists. The two cardiologists will therefore work blind to the examination being evaluated.

SECONDARY OUTCOMES:
Concordance between the diagnosis of TET from perfusion and the 'gold standard' (diagnosis obtained by consensus of two cardiologists based on all blinded examinations of the echo results). Kappa coefficient | visit inclusion
  The two cardiologists will each give their diagnosis independently. If there's a disagreement between them, a third cardiologist (cardiologist number 5) will be called in to help, and the final decision will be made by majority vote.
  The two cardiologists will therefore work blind to the test being evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Yoann MOEUF, medical doctor, Principal Investigator — Hospital Paris Saint-Joseph
Locations (1):
- Hospital Paris Saint-Joseph, Paris, Ilede France, France

IPD SHARING:
Plan to Share IPD: No